CLINICAL TRIAL: NCT01739647
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect on Biomarkers of AZD3293 Including an Open-Label Food Effect Group in Healthy Male and Non-Fertile Female Volunteers
Brief Title: A Single Dose Study to Assess the Safety, Effects, and Blood and Urine Drug Levels of AZD3293 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5010C00001
Record Dates: First submitted 2012-11-30; First posted 2012-12-03 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Young Volunteers; Healthy Elderly Volunteers
Keywords: AZD3293; Healthy volunteers; Elderly volunteers; Phase 1; Single Ascending Dose Study
MeSH Terms: interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD3293 (Experimental): Up to 11 sequential cohorts of healthy young and healthy elderly subjects are planned, with single ascending doses ranging from 1mg to a maximum of 1000mg
  Interventions: Drug: AZD3293
- Placebo (Placebo Comparator): Placebo given (2 subjects in each cohort)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3293 — Oral solution
  Arms: AZD3293
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
This is a single dose study in healthy male and female (of non-child bearing potential) volunteers, to assess the safety, effects on the body, and blood and urine drug levels of AZD3293. AZD3293 is being developed for the treatment of Alzheimer's Disease

DETAILED DESCRIPTION:
A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect on Biomarkers of AZD3293 Including an Open-Label Food Effect Group in Healthy Male and Non-Fertile Female Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) subjects
* Body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* History or presence of psychiatric disease/condition, GI, renal, hepatic, cardiovascular, psychiatric, or retinal diseases or disorders
* History of neurological disease, including seizures, recent memory impairment, or clinically significant head injury
* History of use of antipsychotic drugs , or chronic use of antidepressant or anxiolytic drugs
* Frequent use (more than 2 days per week during the last 12 weeks) of tobacco or other nicotine products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Adverse event monitoring. | From baseline up to 10 days.
Assessment of vital signs and physical examination. | From baseline up to 10 days.
  The vital signs of body temperature, blood pressure and pulse are going to be measured.
Clinical laboratory tests: hematology. | From baseline up to 10 days.
Clinical laboratory tests: urine analysis. | From baseline up to 10 days.
Evaluation of 12-lead digital electrocardiogram (ECG). | From baseline up to 10 days.
  QT/QTc interval, rhythm, rate, morphology is going to be measured.
Assessment of telemetry. | From baseline up to 10 days.
  As reported by investigator.
Columbia-Suicide Severity Rating Scale (C-SSRS) | From baseline up to 10 days.
  Columbia-Suicide Severity Rating Scale (C-SSRS) captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Some questions are yes/no and some are on a scale of 1 (low severity) to 5 (high severity). Completed suicide and non-fatal suicide events are yes/no questions and results presented are the number of participants with these events. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) in the terms of AUC, AUC(0-t), AUC(0-24). | Up 4 days
  Where (AUC(0-t)) is area under the plasma concentration-time curve from zero to the last measurable concentration and (AUC(0-24)) area under the plasma concentration-time curve from zero to 24 hours post-dose.
Investigation on the effect of AZD3293 on biomarkers relevant for Pharmacodynamics in plasma. | Up to 4 days.
  Biomarker PD Aβ (1-40, 1-42) parameters are:
  * Maximum observed plasma concentration (Cmax)
  * Time to Cmax (tmax)
  * Minimum observed plasma concentration (Cmin)
  * Minimum observed plasma concentration below the individual healthy volunteer baseline (pre-dose biomarker concentration prior to dosing) (ΔCmin)
  * Time to Cmin (tmin)
  * Duration (T) of concentration below individual healthy volunteer baseline (BBL), if appropriate for the data (tBBL)
  * Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC(0-t))
  * Area under the plasma concentration-time curve from zero to 24 hours post dose (AUC(0-24))
  * Area under the plasma biomarker concentration curve from time zero to 24 hour that is below individual healthy volunteer baseline (ΔAUC(0-24)).
Investigation of the potential influence of food on Pharmacokinetics (PK) following a single dose of AZD3293. | Up to 4 days.
  Pharmacokinetics (PK) in the terms of plasma Cmax and AUC.
Investigation of the relationship between Pharmacokinetics (PK) and Pharmacodynamics (PD) of AZD3293. | Up to 4 days.
  The Pharmacokinetics (PK) variables may be plasma concentrations or summary measurements such as Cmax or AUC. The Pharmacodynamics (PD) variables may include biomarkers in plasma such as Aβ (1-40, 1-42) or exploratory PD biomarkers, or safety variables.
Pharmacokinetics assessment in the terms of fu (%) (fraction of unbound AZD3293 and AZ13569724 in plasma). | Up to 4 days.
Pharmacokinetics in the terms of Cmax (Maximum observed plasma concentration) and tmax (Time to Cmax ). | Up to 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Alexander, MD, Study Director — AstraZeneca; Ronald Goldwater, MD, Principal Investigator — Parexel
Locations (1):
- Research Site, Baltimore, Maryland, United States